CLINICAL TRIAL: NCT06194110
Title: Comparing the Results of a Stationary and a Mobile Ergospirometry System - a Randomized Crossover Trial
Brief Title: Comparing Stationary and Mobile Ergospirometry
Acronym: QK5_2days
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-16; 2023-01505 (Registry Identifier: EKNZ)
Record Dates: First submitted 2023-12-01; First posted 2024-01-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-08

CONDITIONS: Athletes
Keywords: endurance trained; ergospirometry; Vo2peak

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endurance Trained Athletes
  Interventions: Diagnostic Test: Ergometric test

INTERVENTIONS:
Diagnostic Test: Ergometric test — Ramp test followed by a step test, both with ergospirometry

SUMMARY:
The goal of this randomized crossover trial is to compare the results of a stationary and a mobile ergospirometry system in 20 healthy endurance trained participants. The main question it aims to answer is to investigate the differences in VO2-measurements between the mobile K5 and the stationary Quark ergospirometry system.

Participants will do a maximal ramp test followed by a sub maximal step test with 6 stages on two different days.

DETAILED DESCRIPTION:
20 endurance trained men and/or women will be recruited. A screening will be done before starting with the test protocol on the treadmill to ensure the suitability of the participants. The test protocol includes two parts. The first part is a maximal ramp test (+0.6km/h each minute until exhaustion). The second part includes a step test with 6 sub maximal stages - each lasting 5 minutes - at 50%, 55%, 60%, 70%, 75% and 80% of the maximal velocity achieved in the first part. There will be a short break between the ramp and the step test. The stationary and the mobile system are tested on 2 separate days with a break of 1-3 days in between. On the second day, procedure will be exactly the same for the participants.

ELIGIBILITY:
Inclusion Criteria:

* endurance trained (minimum two times endurance training per week)
* healthy as assessed by the physical-activity-readiness-questionnaire (PAR-Q)
* adequately informed and consent confirmed per signature

Exclusion Criteria:

* Pregnancy based on anamnesis
* acute illness, injury, infection, etc., which would impact the measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy endurance trained male or female older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
VO2 peak | during the last 30 seconds of the ramp test
  Maximal oxygen consumption (VO2) peak values during the ramp test

SECONDARY OUTCOMES:
VO2 | during the last 2 minutes of the step test
  oxygen consumption (VO2) values during step test in steady state
VCO2 | during the last 2 minutes of the step test
  carbon dioxide production (VCO2) values during step test in steady state
Ventilation | during the last 2 minutes of the step test
  Ventilation during step test in steady state
breathing frequency | during the last 2 minutes of the step test
  breathing frequency values during step test in steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No